CLINICAL TRIAL: NCT03002337
Title: Yoga and Aromatherapy on Salivary Hormone and Immune Function in Pregnant Women.
Brief Title: Efficacy of the Yoga and Aromatherapy on Salivary Hormone and Immune Function in Pregnant Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Pao-Ju chen, Principal Investigator, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2-102-05-148
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Stress, Psychologic
Keywords: aromatherapy massage, yoga
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aromatherapy massage (Experimental): Ten aromatherapy group received 70 minutes of aromatherapy massage once biweekly by certified aromatherapy therapist for 20 weeks.
  Interventions: Behavioral: Aromatherapy massage
- Yoga exercise (Experimental): The yoga group participated in two weekly 70-minute yoga sessions led by a midwife certified as a yoga instructor for 20 weeks
  Interventions: Behavioral: Yoga exercise
- Control (No Intervention): the control group received only routine prenatal care.

INTERVENTIONS:
Behavioral: Aromatherapy massage — All of the participants in the aromatherapy group underwent aromatherapy massage for 70 minutes every two weeks between 16 to 36 weeks GA (ten sessions total). The aromatic massage oils were composed of 2 c.c. lavender (Lavandula angustifolia) blended with 98 c.c. almond oil. This concentration of the mixed essential oil was kept at room temperature for massage use.
  Arms: Aromatherapy massage
Behavioral: Yoga exercise — Prenatal yoga was offered in six 70-minute yoga sessions per week for 20 weeks, with 10-12 women in each session. Each participant should attend two sessions of yoga every two days, held in a quiet room near the prenatal clinic. Yoga specifically designed for women during the second and third trimesters, was guided by a midwife who was certified as a yoga instructor. Yoga included physical postures/ stretch, deep breathing, guided imagery, and deep relaxation. Before each posture/stretch, the instructor guided participants to relax each body part and calm their mind.
  Arms: Yoga exercise

SUMMARY:
This study's aims are to examine the effects of yoga and aromatherapy on women's stress and immune function during pregnancy.

DETAILED DESCRIPTION:
This longitudinal, prospective, randomized controlled trial recruited 75 healthy pregnant women from a prenatal clinic in Taipei using convenience sampling. The participants were randomly assigned to the aromatherapy group (n=25), yoga group (n=25) or control (n=25) group using Clinstat block randomization.

The aromatherapy group received 70 minutes of aromatherapy massage once biweekly for 20 weeks; the yoga group participated in two weekly 70-minute yoga sessions led by a midwife certified as a yoga instructor for 20 weeks; the control group received only routine prenatal care. All participants' salivary cortisol and immunoglobulin A levels were collected before and after yoga or aromatherapy every 4 weeks from 16 to 36 weeks' gestation.

To collect a sufficient quantity of saliva, we used Salivette® cotton swabs (Salimetrics, State College, PA, USA), which were stored in double-layer plastic tubes with a lid. When participants chew a swab for about 2 to 3 minutes, saliva flow is stimulated to a sufficient amount (1 mL) for collection. After the tube was centrifuged at 1000 x g for 2 minutes, saliva was stored at -80°C until assay for salivary cortisol and IgA concentrations.

Cortisol was measured using a competitive enzyme-linked immunoassay (ELISA) kit (Cayman Chemical Company, USA), and salivary IgA was measured using double-antibody sandwich ELISA method per the manufacturer's instruction (ICL, Inc., USA).

ELIGIBILITY:
Inclusion Criteria:

* Normal pregnancy
* Age 20-45 years
* Agreed to follow-up collections of saliva samples
* Could read and write Chinese

Exclusion Criteria:

* Oral steroid use
* History of severe illness (e.g., heart disease, systemic lupus erythaematosus, metabolic disorders) or depression.
* Drug use (prescribed or illicit).
* High-risk pregnancy (i.e., first-trimester vaginal bleeding, artificially insemination, multiple gestations, foetal growth restriction or other abnormalities).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Physiological parameter (salivary cortisol) | 20 weeks
  This study used salivary cortisol as the indicator of stress. To assess stress in this study, the concentrations of cortisol (μg/dL) in saliva samples were analysed and was measured using a competitive enzyme-linked immunoassay (ELISA) kit (Cayman Chemical, Ann Arbor, USA). The participants' salivary cortisol levels were collected before and after the intervention group received aromatherapy massage (every month from 16 to 36 weeks gestation).

SECONDARY OUTCOMES:
Physiological parameter (salivary IgA) | 20 weeks
  This study used salivary IgA as the indicator of immune function. To assess immune function in this study, the concentrations of IgA (μg/mL) in saliva samples were analysed and was measured using the double-antibody sandwich ELISA method according to the manufacturer's instructions (ICL, Inc., USA). The participants' salivary immunoglobulin A levels were collected before and after the intervention group received aromatherapy massage (every month from 16 to 36 weeks gestation).

IPD SHARING:
Plan to Share IPD: No